CLINICAL TRIAL: NCT06236061
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Active-controlled Study to Evaluate the Efficacy and Safety of LCZ696/Amlodipine 200/2.5 mg, 200/5 mg and 200/10 mg Compared to LCZ696 200 mg Alone in Patients With Grade 1 and 2 Hypertension Not Adequately Controlled by LCZ696 200 mg Monotherapy
Brief Title: Study of Efficacy and Safety of LCZ696/Amlodipine in Grade 1 and 2 Hypertension Patients Uncontrolled by LCZ696 Monotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLAZ696B11302
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Hypertension
Keywords: LCZ696; Phase 3; grade 1 and 2 hypertension; Amlodipine
MeSH Terms: conditions — Hypertension; Lymphoma, Follicular | interventions — sacubitril and valsartan sodium hydrate drug combination; Amlodipine

STUDY DESIGN:
Intervention Model Description: This study is composed of two parts; the Core part including double-blind period, and the open-label extension (OLE) part.
  The Core part is a parallel model, and the OLE is a sequential model.
Who Masked: Participant, Care Provider, Investigator
Masking Description: In the Core part, Participant, care provider and Investigator will be masked. In the OLE part, no masking to anyone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LCZ 200mg (Active Comparator): Oral administration, 1 tablet of LCZ 200 mg daily, 4 capsules of Amlodipine placebo daily.
  Interventions: Drug: LCZ; Other: Placebo
- LCZ 200mg + AML 2.5mg (Experimental): Oral administration, 1 tablet of LCZ 200 mg daily, 1 capsule of Amlodipine 2.5 mg daily and 3 capsules of Amlodipine placebo daily.
  Interventions: Drug: LCZ/AML 200 mg/2.5 mg; Other: Placebo
- LCZ 200mg + AML 5mg (Experimental): Oral administration, 1 tablet of LCZ 200 mg daily, 2 capsules of Amlodipine 2.5 mg daily and 2 capsules of Amlodipine placebo daily.
  Interventions: Drug: LCZ/AML 200 mg/5 mg; Other: Placebo
- LCZ 200mg + AML 10mg (Experimental): Oral administration, 1 tablet of LCZ 200 mg daily, 4 capsules of Amlodipine 2.5 mg daily.
  Interventions: Drug: LCZ/AML 200 mg/10 mg

INTERVENTIONS:
Drug: LCZ — LCZ 200 mg
  Other Names: LCZ696
  Arms: LCZ 200mg
Drug: LCZ/AML 200 mg/2.5 mg — LCZ/AML 200 mg/2.5 mg
  Other Names: LCZ696/Amlodipine
  Arms: LCZ 200mg + AML 2.5mg
Drug: LCZ/AML 200 mg/5 mg — LCZ/AML 200 mg/5 mg
  Other Names: LCZ696/Amlodipine
  Arms: LCZ 200mg + AML 5mg
Drug: LCZ/AML 200 mg/10 mg — LCZ/AML 200 mg/10 mg
  Other Names: LCZ696/Amlodipine
  Arms: LCZ 200mg + AML 10mg
Other: Placebo — Matching placebo of Amlodipine.
  Arms: LCZ 200mg; LCZ 200mg + AML 2.5mg; LCZ 200mg + AML 5mg

SUMMARY:
This CLAZ696B11302 study is composed of two parts; the Core part including double-blind period, and the open-label extension (OLE) part which is an open-label extension of the Core part.

The purpose of the Core part is to demonstrate that LCZ696 (LCZ) when used in combination with amlodipine (AML), denoted as LCZ/AML, will provide greater blood pressure lowering benefit compared to LCZ monotherapy in patients with grade 1 and 2 hypertension not adequately controlled with LCZ monotherapy. The purpose of the OLE part is to assess the long-term safety, tolerability and efficacy of the treatment with LCZ/AML.

DETAILED DESCRIPTION:
This study is designed to provide efficacy and safety data for combinations of LCZ 200 mg and AML (2.5 mg, 5 mg or 10 mg) as compared to LCZ monotherapy in patients with grade 1 and 2 hypertension not adequately controlled with LCZ monotherapy, and also the long-term safety, tolerability and efficacy of the treatment with LCZ/AML. The Core part is a multicenter, randomized, double-blind, parallel-group, active-controlled study which is comprised of the following three periods: Screening / washout period, Single-blind active run-in period, Double-blind treatment period (8 weeks). A 52 week, open-label extension part will be conducted following the completion of the Core part. Those participants that complete the Core part without permanent study drug discontinuation will be offered continued participation in an additional 1 year safety extension to the protocol. Of the patients completed the Core part, approximately 278 participants who are eligible and agree to participate and sign a new informed consent form will start the OLE part, and receive the open-label LCZ/AML combination drug through the OLE part. At start of the OLE part, all participants will be switched to the open-label LCZ/AML 200 mg/5 mg combination drug from double-blinded study medication. After 4 weeks of OLE part, the dosage will be titrated up to LCZ/AML 200 mg/10 mg if an adequate control in blood pressure is not achieved [msSBP ≥ 130 mmHg or msDBP ≥ 80 mmHg, or the Investigator's judgement basically in accordance with the current local hypertension treatment guideline (JSH2019)] and when there is no safety concern on up-titration judged by the Investigator. If the blood pressure is controlled optimally, the participants will continue to receive LCZ/AML 200 mg/5 mg. Down-titration from LCZ/AML 200 mg/5 mg to LCZ/AML 200 mg/2.5 mg is permitted after the start of OLE part if participants are having difficulty with the current treatment of LCZ/AML 200 mg/5 mg due to adverse events (AEs) etc. Dose adjustment (up or down-titration) is allowed if participants meet the criteria for dose adjustment (the same defined above as up-titration and down-titration). The Investigators should maintain the maximum tolerated dose as much as possible after 8 weeks of OLE part. Thiazide diuretics/thiazide-like diuretics are allowed as rescue medication(s) at the investigator's discretion on and after 8 weeks of OLE part, if blood pressure is not adequately controlled even with LCZ/AML 200 mg/10 mg or maximum tolerated dose and with no signs of hypovolemia. Initial dose of the concomitant diuretics should be low, then the dose can be adjusted.

ELIGIBILITY:
Inclusion Criteria:

Core Part)

* Patients with grade 1 and 2 essential hypertension, untreated or currently taking antihypertensive therapy

  1. Untreated patients [either newly diagnosed with essential hypertension or those with a history of hypertension but have not been taking any antihypertensive drugs for 4 weeks prior to screening visit (Visit Scr)] must have a msSBP of ≥ 150 mmHg and < 180 mmHg at both screening (Visit Scr) and run-in visit (Visit Run-in)
  2. Pretreated patients (taking antihypertensive drugs within 4 weeks prior to screening visit (Visit Scr)) must have msSBP < 180 mmHg at screening visit (Visit Scr), and msSBP ≥ 150 mmHg and < 180 mmHg at run-in visit (Visit Run-in)
* Patients who are not adequately responsive to LCZ 200 mg treatment must have a msSBP ≥ 140 mmHg and < 180 mmHg at the end of run-in/randomization visit
* Patients who are able to communicate well with the Investigator, to understand and comply with all study requirements, and demonstrate good medication compliance (≥ 80% compliance rate) during the single-blind run-in period OLE part)
* Patients who have completed the Core part without permanent study drug discontinuation and who, as judged by the Investigator, are able to continue in the OLE part
* Patients who have msSBP < 160 mmHg and msDBP <100 mmHg at Visit W8 of the double-blind period

Exclusion Criteria:

Core part)

* Patients currently on one or more antihypertensive medications in whom the Investigator considers that the medications cannot be safely discontinued for the duration of the Core part
* Severe hypertension (msSBP ≥ 180 mmHg and/or msDBP ≥ 110 mmHg at any visit prior to or at randomization), or malignant hypertension
* History or evidence of a secondary form of hypertension, including but not limited to any of the following: renal parenchymal hypertension, renovascular hypertension (unilateral or bilateral renal artery stenosis), coarctation of the aorta, primary hyperaldosteronism, Cushing's disease, pheochromocytoma, polycystic kidney disease, sleep apnea, and drug-induced hypertension
* Patients with Type 1 or Type 2 diabetes mellitus not well controlled based on the Investigator's clinical judgement
* Concomitant refractory angina pectoris [angina in setting of Coronary Artery Disease (CAD) which is uncontrolled by combination of optimal medical therapy, angioplasty or bypass surgery]
* Clinically significant valvular heart disease at screening
* Any history of stroke or hypertensive encephalopathy
* History of hypersensitivity to any of the study treatments or its excipients, ARBs or to drugs of similar chemical classes
* Use of other investigational drugs within 30 days or 5 half-lives of screening visit, whichever is longer OLE part)
* Any medical condition that in the opinion of the Investigator is likely to prevent the patient from safely tolerating LCZ/AML or complying with the requirements of the study
* Patients who have experience of angioedema event(s) which occurred and reported by the Investigator during the Core part of study
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 10 days after stopping study treatment. Highly effective contraception methods are defined as same as the criteria for the Core part.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
[Core Part] Change from baseline to Week 8 in msSBP | Baseline, Week 8
  Change from baseline to Week 8 in mean sitting systolic blood pressure (msSBP)

SECONDARY OUTCOMES:
[Core Part] Change from baseline to Week 8 in maSBP | Baseline, Week 8
  Change from baseline to Week 8 in mean 24-hour ambulatory systolic blood pressure (maSBP)
[Core Part] Proportion of patients achieving a blood pressure control after 8 weeks of treatment | 8 weeks
  Proportion of patients achieving a blood pressure control (msSBP <140 mmHg and msDBP <90 mmHg) after 8 weeks of treatment
[Core Part] Change from baseline to Week 8 in msDBP | Baseline, Week 8
  Change from baseline to Week 8 in mean sitting diastolic blood pressure (msDBP)
[Core Part] Change from baseline to Week 8 in maDBP | Baseline, Week 8
  Change from baseline to Week 8 in mean 24-hour ambulatory diastolic blood pressure (maDBP)
[Core Part] Proportion of patients achieving a msSBP response after 8 weeks of treatment | 8 weeks
  Proportion of patients achieving a msSBP response (<140 mmHg or a reduction ≥20 mmHg from baseline) after 8 weeks of treatment
[Core Part] Proportion of patients achieving a msDBP response after 8 weeks of treatment | 8 weeks
  Proportion of patients achieving a msDBP response (<90 mmHg or a reduction ≥10 mmHg from baseline) after 8 weeks of treatment
[Core Part] Change from baseline to Week 8 in daytime, nighttime and early morning maSBP | Baseline, Week 8
  Change from baseline to Week 8 in daytime, nighttime and early morning maSBP
[Core Part] Change from baseline to Week 8 in daytime, nighttime and early morning maDBP | Baseline, Week 8
  Change from baseline to Week 8 in daytime, nighttime and early morning maDBP
[Core Part] Number of patients with treatment-emergent adverse events | Up to 8 weeks
  Number of patients experiencing treatment-emergent adverse events including (but not limited to) any unfavorable and unintended signs, symptoms or disease, abnormal vital signs, electrocardiogram data, safety lab measurements that induce clinical signs or symptoms, are considered clinically significant or require therapy
[OLE Part] Number of patients with treatment-emergent adverse events | Up to 52 weeks
  Number of patients experiencing treatment-emergent adverse events including (but not limited to) any unfavorable and unintended signs, symptoms or disease, abnormal vital signs, electrocardiogram data, safety lab measurements that induce clinical signs or symptoms, are considered clinically significant or require therapy
[OLE Part] Change from baseline in msSBP and msDBP | Baseline, Week 4, Week 8, Week 13, Week 26, Week 39, and Week 52 of OLE part
  Change from baseline in msSBP and msDBP by visit in OLE part
[OLE Part] Proportion of patients achieving blood pressure control, msSBP response and msDBP response | Over 52 weeks
  Proportion of patients achieving blood pressure control (msSBP <140 mmHg and msDBP <90 mmHg), msSBP response (<140 mmHg or a reduction ≥20 mmHg from baseline) and msDBP response (<90 mmHg or a reduction ≥10 mmHg from baseline) by visit

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- Japan (32):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Itoshima, Fukuoka
  - Novartis Investigative Site, Chitose, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kamakura, Kanagawa
  - Novartis Investigative Site, Kawasaki-shi, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Ōsaki, Miyagi
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Chiyoda City, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Musashino, Tokyo
  - Novartis Investigative Site, Nerima Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Shinagawa-Ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Suginami-ku, Tokyo
  - Novartis Investigative Site, Toshima-Ku, Tokyo
  - Novartis Investigative Site, Chuoh-ku
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com